CLINICAL TRIAL: NCT05204849
Title: Use of ACTIVE Fluid Exchange to Treat Intraventricular Hemorrhage
Brief Title: ACTIVE Study - Use of ACTIVE Fluid Exchange to Treat Intraventricular Hemorrhage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); IRRAS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 47723569
Record Dates: First submitted 2021-12-15; First posted 2022-01-24 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2021-12

CONDITIONS: Intraventricular Hemorrhage
Keywords: Intraventricular Hemorrhage; Ventriculostomy; Catheter occlusions; Catheter-Related Infections; Clearance of blood; Active irrigation and aspiration; IRRAflow
MeSH Terms: conditions — Catheter-Related Infections

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial, 1:1 fashion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active irrigation and aspiration (Active Comparator): Patients randomized to IRRAflow will receive a ventricular catheter with active irrigation and aspiration.
  Interventions: Device: IRRAflow
- Standard passive external ventricular drainage (Active Comparator): Patients randomized to passive external ventricular drainage will receive a standard EVD.
  Interventions: Procedure: Standard ventriculostomy

INTERVENTIONS:
Device: IRRAflow — Ventriculostomy using IRRAflow with active irrigation and aspiration
  Arms: Active irrigation and aspiration
Procedure: Standard ventriculostomy — Standard passive external ventricular drainage
  Arms: Standard passive external ventricular drainage

SUMMARY:
Randomised controlled trial evaluating active irrigation using IRRAflow device in patients with intraventricular hemorrhages (IVH). Patients will be randomized in a 1:1 fashion to IRRAflow active irrigation and aspiration compared to standard passive external ventricular drainage.

The investigators hypothesize that active irrigation using the IRRAflow system will reduce the occlusion rates of the ventricular drain. Further, reduce the rate of catheter related infection and reduce time needed for clearance of blood from the intraventricular space compared with passive drainage alone. Further more, reduce treatment time, patient length of stay, and overall treatment cost when compared with passive drainage.

DETAILED DESCRIPTION:
Intraventricular extension of hemorrhage (IVH) is a particularly poor prognostic sign, with expected mortality between 50% and 80%. IVH is a significant and independent contributor to morbidity and mortality, yet therapy directed at ameliorating intraventricular clot has been limited. Conventional therapy centers on managing hypertension and intracranial pressure while correcting coagulopathy and avoiding complications such as rebleeding and hydrocephalus. Surgical therapy alone has not changed the natural history of the disease significantly. Although ventriculostomy appears to be effective in controlling ICP, this technique does little to reduce morbidity and does not address the inflammatory process. The severity of communicating hydrocephalus appears to be related to IVH volume and the duration of exposure of CSF to clotted blood.

Management of hemorrhagic patients is typically orchestrated by neurosurgeons and neuro-intensivists. Comprehensive care should include surveillance and monitoring of intracranial pressure (ICP), Cerebral Perfusion Pressure (CPP), and hemodynamic function. Furthermore, prevention of infection, complications of immobility through positioning and mobilization within physiological tolerance play an important role in optimizing outcomes after intracerebral hemorrhage (ICH).

There are multiple approaches to facilitating Cerebrospinal Fluid (CSF) drainage and intracranial pressure (ICP) monitoring. Routinely, ICP is measured by use of devices inserted into the brain parenchyma or cerebral ventricles. A Ventricular Catheter (VC) inserted into the lateral ventricle allows for drainage of CSF to help reduce ICP.

The IRRAflow system performs active, controlled fluid exchange, based on the notion that it is faster to wash out IVH, compared to gravity drainage alone. IRRAflow combines periodic, controlled irrigation and aspiration of the catheter probe with neutral physiological fluids. The continuous perfusion cleans the entire inner catheter probe's surface while the fluid movement helps to disrupt potential clot or bacteria colony formation on the catheter probe's intracranial external surface, thereby eliminating the underlying reasons for the problems associated with passive drainage: blockage and infection. Furthermore, IRRAflow perfusion is combined with continuous ICP monitoring that includes safety alarms. Contrary, with passive drainage, such as today's standard of care, the external ventricular drain (EVD), is inherently inefficient because of its inability to overcome blood clot adhesion. As a result, EVD's generally need a lot of treatment time for the evacuation of a clinically significant blood volume and often leave enough volume of residual blood to create secondary adverse effects, like hydrocephalus. IRRAflow was designed to increase drainage efficiency by means of gradual and continuous dilution of the pathological intracranial fluids through irrigating the catheter with physiological fluids as well as the continuous pressure fluctuations inside the pathological collection, which are created by the appropriate irrigation patterns. By design, the IRRAflow catheter probe is irrigated regularly in a way that maintains its patency. Catheter blockages are theoretically very unlikely since any material build-up at the catheter's tip is washed away during the next irrigation phase, which will occur in, at most, a couple of minutes. Additionally, the volume and flow rate of each irrigation is such that the length of the IRRAflow catheter probe's outer surface is washed by backflow, thus arguably reducing the chance for bacterial colonisation (Data on File at IRRAS). As for safety, IRRAflow automatically, reliably, and continuously monitors ICP and alerts hospital personnel with visual and sound alarms immediately when the patient's ICP is out of the pressure range set by the treating neurosurgeon, which eliminates any delay in detecting under or over drainage and any treatment's compromise.

The clinical efficacy of the IRRAflow system is currently validated to a limited extent based on case series (Evidence grade 4) with a total number of patients around 200 distributed across multiple countries including in Greece, India, Sweden, Germany, UK, USA, and Finland. The system has been used to treat subarachnoid, intraventricular, intraparenchymal, and subdural hemorrhages. The system was CE Marked in 2014 and began limited market release in Germany in 2017. It received US FDA clearance in July of 2018 and began to be used commercially based on the conclusion that the device was safe. Case report data on the 200 initial patients has been collected by the company and maintained on file. The data has shown that zero IRRAflow catheter occlusions have been experienced when the irrigation setting has been activated (unpublished). Furthermore, treatment times were much shorter and posttreatment residual blood volumes were less than expected by the treating neurosurgeons (31), (Data on File at IRRAS). To date there have not been any documented blockages or probe associated infections detected in any IRRAflow treatment.

At present time, there is no level 1 evidence for treatment efficacy. However, the treatment is new and intuitively rational, and it is applied for patients with intraventricular hemorrhage, which has an extremely high mortality and morbidity rate, for whom there are no other treatment options.

In light of the above, the current clinical ACTIVE study is being initiated to evaluate the hypothesis that active irrigation by IRRAflow® will reduce the time needed for clearance of intraventricular blood from intraventricular space compared with passive drainage. Further, active controlled irrigation can improve catheter occlusion and infection rates compared with passive drainage. This is accomplished through IRRAflow's mechanism of action, Active Fluid Exchange (continuous, intelligent irrigation combined with continuous drainage and ICP monitoring). This active fluid exchange could enable an optimal washout of the ventricles thus leading to better outcomes than traditional treatment. Clinical evidence supporting this hypothesis has already been established by Zhang et al., 2007, and the aforementioned article. The investigators aim to provide that similar results can be obtain through less invasive methods.

The investigators expect that the ACTIVE study will provide the first grade 1 evidence to date characterizing the IRRAflow IVH clearance performance, documenting device safety, and additionally provide preliminary indications of the potential correlated improvements in clinical outcome and cost-effectiveness of treatment as well as a potential reduction in post-surgical complications such as post-ictus hydrocephalus and central nervous system (CNS) infection. Endpoints and objectives are elaborated further below. If positive, the Study will provide a pivotal argument for the use of active fluid exchange in the treatment of hemorrhagic stroke with ventricular involvement, potentially changing standard practice for the better

The proposed study is a multi center prospective, controlled, randomized trial to evaluate the efficacy and safety of evacuation of intraventricular hematoma by Active external ventricular drainage (INTERVENTION - IRRAflow) compared to passive external ventricular drainage (CONTROL - EVD).

Randomization of the study will occur following enrollment upon the patient presentation to the emergency room. Upon initial diagnosis and enrollment, if it is determined that a CSF drainage is necessary, the patient will be randomized to either the IRRAflow with Active Fluid Exchange arm (intervention) or a standard practice EVD arm (control). The randomization will occur in a 1 to 1 fashion. This means, that 50% of cases will be randomized to the intervention and 50% to control. Drainage therapy with EVD or IRRAflow will commence for as long as it is deemed necessary by the treating physician. All patients enrolled in the trial will receive additional supportive and medical treatment by choice of the treating physician and in accordance with standard of care. Such treatment may include neurointensive care, neuromonitoring, and surgical or endovascular occlusion identified sources of intracranial hemorrhage, e.g. vascular anomalies, aneurisms, etc. Interventional treatment will be stopped in case of 1) patient exclusion from the trial, 2) ethical or medical safety contraindications for further interventional treatment determined by the Investigators.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years of age
2. Intraventricular hemorrhage documented on head CT or MRI scan, no older than 24 hrs.
3. Intraventricular hemorrhage Graeb Score ≥3 points
4. Urgent need of cerebrospinal fluid drainage (<24 hours)
5. Deterioration of consciousness or medical sedation at the time of enrollment causing the patient to be mentally and/or physically incapacitated and legally incompetent in the decision of inclusion ("acute study" conduct).
6. Indication for active treatment evaluated by the treating physicians
7. Use of validated anti-conception in fertile female participants in concordance with guidelines provided by the Danish Health and Medicines Authority or a negative urine human chorion gonadotropin (HCG) test.

Exclusion Criteria:

1. Patient has fixed and dilated pupils
2. Pregnant or nursing women (fertile female participants will be required to take a validated pregnancy test for evaluation of pregnancy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2022-01-13 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Drain survival time | Time with ventricular catheter from placement to fist observed occlusion, an average of 11 days
  Time to first observed occlusion of the catheter

SECONDARY OUTCOMES:
Catheter related infections | Time with ventricular catheter from placement to fist observed occlusion, an average of 11 days
  Rate of ventriculitis and meningitis related to the ventriculostomy
Rate of shunt dependency | During the first 90 days after intervention
  No. of patients with resistent need of CSF drainage receiving a ventriculo-peritoneal (VP)-shunt
Time to clearance of blood | At day 0, 2, 4, 6, 8
  CT volume of head CT scans
Length of stay at the ICU | Expected between 1 and 30 days
  Length of stay at the ICU
Functional outcomes - eGOS and mRS | At inclusion, at discharge (an average of 30 days) and 90 days
  Extended glasgow outcome scale and modified rankin scale
Mortality rate | At 30 days and 90 days
  Evaluation of mortality rates

CONTACTS AND LOCATIONS:
Overall Officials: Anders Korshøj, MD, PhD, Principal Investigator — Dept. of Neurosurgery, Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Protocol will be published primo 2022.

REFERENCES:
- [Derived] Haldrup M, Rasmussen M, Mohamad N, Dyrskog S, Thorup L, Mikic N, Wismann J, Gronhoj M, Poulsen FR, Nazari M, Rehman NU, Simonsen CZ, Korshoj AR. Intraventricular Lavage vs External Ventricular Drainage for Intraventricular Hemorrhage: A Randomized Clinical Trial. JAMA Netw Open. 2023 Oct 2;6(10):e2335247. doi: 10.1001/jamanetworkopen.2023.35247. PMID 37815832
- [Derived] Haldrup M, Mohamad N, Rasmussen M, Thorup L, Dyrskog S, Simonsen CZ, Miscov R, Bjarkam CR, Gronhoj M, Poulsen FR, Korshoj AR. Study protocol for ACTIVE study: safety and feasibility evaluation of external ventricular drainage with ACTIVE fluid exchange in intraventricular hemorrhage-a phase 2, multi-center, randomized controlled trial. Trials. 2022 Dec 29;23(1):1062. doi: 10.1186/s13063-022-07043-9. PMID 36581996